CLINICAL TRIAL: NCT03197779
Title: A Randomized, Double-Blind, Placebo-Controlled, Ascending-Dose Short and Long Intravenous Infusion Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of BMS- 962212 in Healthy Subjects
Brief Title: A Short and Long Intravenous Infusion Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of BMS-962212 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV001-001
Record Dates: First submitted 2017-06-21; First posted 2017-06-23 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Thrombosis
MeSH Terms: conditions — Thrombosis | interventions — BMS-962212; Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- BMS-962212 Two Hour Administration (Experimental): Intravenous administered over 2 hours of BMS-962212
  Interventions: Drug: BMS-962212
- BMS-962212 5 Day Administration (Experimental): Intravenous administered over 5 days of BMS-962212
  Interventions: Drug: BMS-962212
- BMS-962212 and Aspirin (Experimental): BMS-962212 intravenous administration, followed by aspirin oral administration, then combination administration of BMS-962212 and aspirin
  Interventions: Drug: BMS-962212; Drug: Aspirin
- Placebo and Aspirin (Placebo Comparator): Placebo intravenous administration, followed by aspirin, then combination administration of placebo and aspirin
  Interventions: Drug: Aspirin; Other: Placebo
- Placebo (Placebo Comparator): Placebo intravenous administration
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BMS-962212 — Intravenous Infusion administration over 2 hours or 5 days
  Arms: BMS-962212 5 Day Administration; BMS-962212 Two Hour Administration; BMS-962212 and Aspirin
Drug: Aspirin — Oral administration
  Arms: BMS-962212 and Aspirin; Placebo and Aspirin
Other: Placebo — Oral administration
  Arms: Placebo; Placebo and Aspirin

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics following increasing doses of 2 h (Part A) and 5 day (Part B) continuous IV infusions of BMS-962212 in healthy subjects across the expected pharmacodynamic dose range.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examination, ECG, and clinical laboratory determinations
* Body Mass Index (BMI) of 18 to 32 kg/m2 inclusive [as calculated by BMI = weight (kg)/ [height (m)]2
* This study permits the re-enrollment of a subject that has discontinued the study as a pre-treatment failure (ie, subject has not been randomized / has not been treated). If re-enrolled, the subject must be re-consented
* Men, ages 18 to 45 years, inclusive; women, ages 18-45, who are not of child-bearing potential
* Women must not be breastfeeding

Exclusion Criteria:

* Any significant acute or chronic medical illness
* Women of child-bearing potential
* Current or recent (within 3 months of study drug administration) gastrointestinal disease which by the judgment of the Investigator may increase a subject's risk of gastrointestinal bleeding (e.g., peptic or gastric ulcer disease, severe gastritis, history of gastrectomy)
* Any major surgery within 12 weeks of study drug administration
* History of blood transfusion, clinically significant bleeding event(s), or documented genetic bleeding diathesis or thrombophilia
* For Aspirin Containing Arm Participants Only: Known allergy to non-steroidal anti-inflammatory drugs or history of intolerance or abnormal sensitivity to aspirin (e.g gastrointestinal intolerance, bruising or bleeding, aspirin induced breathing difficulties or nasal polyps)

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 691 (Actual)
Dates: Start 2013-11-18 (Actual); Primary Completion 2016-02-02 (Actual); Study Completion 2017-01-24 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AE) | Up to 8 days
  measured by incidence
Serious Adverse Events (SAE) | Up to 8 days
  measured by incidence
Discontinuation due to AE | Up to 8 days
  measured by incidence
Death | Up to 8 days
  measured by incidence
AE of clinically significant bleeding | Up to 8 days
  measured by incidence
AE of clinically significant infusion reaction | Up to 8 days
  measured by incidence
AE of clinically significant vital signs | Up to 8 days
  measured by incidence
QTcF intervals - QT interval corrected for heart rate according to Fridericia's formula | Up to 8 days
  measured by ECG
QRS - The interval from the beginning of the Q wave and the end of the S wave | Up to 8 days
  measured by ECG
PR - The interval from the beginning of the P wave to the beginning of the QRS complex | Up to 8 days
  measured by ECG
24-hour cardiac monitoring | Up to 6 days
  measured by telemetry
Glomerular filtration rate (GFR) | Up to 8 days
  measured by iohexol administration plasma clearance and the Chronic Kidney Disease-Epidemiology Collaborative Group (CKD EPI) equation
Cystatin-C | Up to 8 days
  measured by serum biomarkers
Neutrophil gelatinase-associated lipocalin (NGAL) | Up to 8 days
  measured by urine biomarkers
Monocyte chemoattractant protein-1 (MCP-1) | Up to 8 days
  measured by urine biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - Wcct Global, Llc, Cypress, California
  - California Clinical Trials Medical Group, Glendale, California
  - Parexel International - Baltimore Epcu, Baltimore, Maryland

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx